CLINICAL TRIAL: NCT04764552
Title: Effect of Yeahhh Baby! Ointment on Efficacy to Relieve Joint Pain in Men and Women With Hip and/or Knee Pain
Brief Title: Yeahhh Baby! Ointment on Hip and/or Knee Pain in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: YEAHHH! BABY LLC (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2021-94
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Joint Pain
Keywords: hip; knee; topical
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Intervention Model Description: double-blinded crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yeahhh Baby Ointment (Experimental): Ointment will be applied per instructions twice daily during treatment with a two week washout period between arms.
  Interventions: Dietary Supplement: Yeahhh Baby Ointment
- Placebo Ointment (Placebo Comparator): Ointment will be applied per instructions twice daily during treatment with a two week washout period between arms.
  Interventions: Other: Coconut oil ointment

INTERVENTIONS:
Dietary Supplement: Yeahhh Baby Ointment — The ointment consists primarily of coconut oil (98%), with small amounts of herbal ingredients (tanner's bark, slippery root, sweet weed, velvet plant, walnut hulls, kidney root, green ginger, Indian pink, mad dogweed, and nigella seed) thought to reduce inflammation and to promote tissue healing.
  Arms: Yeahhh Baby Ointment
Other: Coconut oil ointment — Coconut oil ointment with a little olive oil.
  Arms: Placebo Ointment

SUMMARY:
This study will compare the impact of the Yeahhh Baby! Ointment, as compared to a placebo, on measures of joint pain and discomfort in those who regularly experience joint pain. The hypothesis is that perceived pain will be reduced when subjects use the Yeahhh Baby! Ointment. Previous studies exploring the efficacy of topicals on joint pain relief have used a similar design and similar joint pain assessments as employed herein (The Western Ontario and McMaster Universities Arthritis Index [WOMAC] and visual analog scale [VAS] for pain).

DETAILED DESCRIPTION:
Joint pain is a common ailment among adults in the United States. In 2014, an estimated 14.6 million Americans with arthritis suffered from severe joint pain. It is therefore unsurprising that many topical ointments are currently marketed for joint pain relief including Bengay®, Icy Hot®, Jointflex®, and Aspercreme®. These ointments aim to reduce pain often through a combination of analgesic ingredients include capsaicin, salicylates, menthol, camphor, and lidocaine. Bengay® products, for instance, contain one or more of menthol, camphor, salicylates, and lidocaine. Icy Hot® products contain menthol, while some also include lidocaine.

Yeahhh Baby! ointment is an herbal (botanical: plant-based) treatment for those impacted by joint pain. The product contains a variety of herbal ingredients that have been touted by some within the alternative medicine community as "healing agents." The product started selling in 2016 and is available commercially as an all-natural alternative to other commercially available products. This ointment consists primarily of coconut oil (98%), with magnesium and small amounts of herbal ingredients (tanner's bark, slippery root, sweet weed, velvet plant, walnut hulls, kidney root, green ginger, Indian pink, mad dogweed, and nigella seed) thought to reduce inflammation and to promote tissue healing.

The present study will compare the impact of the Yeahhh Baby! Ointment, as compared to a placebo, on measures of joint pain and discomfort in those who regularly experience joint pain. The hypothesis is that perceived pain will be reduced when subjects use the Yeahhh Baby! Ointment. Previous studies exploring the efficacy of topicals on joint pain relief have used a similar design and similar joint pain assessments as employed herein (The Western Ontario and McMaster Universities Arthritis Index [WOMAC] and visual analog scale [VAS] for pain).

ELIGIBILITY:
Inclusion Criteria:

* Self-reported joint pain with a minimum pain rating of 3/10 for at least the past 30 days
* Recreationally active (2 or more days per week)
* Not obese (BMI < 30kg/m2)

Exclusion Criteria:

* Tobacco users/Smokers
* Allergic to coconut, walnuts, oak, olives
* Currently using anti-inflammatory medicines or dietary supplements (and not willing to cease for one-month prior to participation and throughout study)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Joint pain visual analog scale | days 1-14
  A 100mm visual analog scale will be used to assess join pain. Scores range from 0 (subject strongly disagreeing with prompt) to 100 (strongly agree)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | days 1-14
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68) with 0 being none and high values being most.
Blood pressure | First 1 day
  Resting blood pressure will be measured.
Blood pressure | 15th day
  Resting blood pressure will be measured.
Heart Rate | First 1 day
  Resting heart rate will be measured.
Heart Rate | 15th day
  Resting heart rate will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Reseach, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No